CLINICAL TRIAL: NCT03204448
Title: Evaluation of Clinical Performance of Serologic Anti-Ro60 Autoantibody Detection Kit on BioCLIA Platform
Brief Title: Clinical Performance of BioCLIA Ro60
Status: Withdrawn | Type: Observational
Why Stopped: Evaluation halted
Sponsor: HOB Biotech Group (Industry)
Responsible Party: Sponsor
Other Study IDs: CRM CSP 001
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Systemic Lupus Erythematosus; Sjogren's Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Clinically leftover plasma/serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Relevant Disease Samples: Samples are tested on BioCLIA Ro60 instrument with Ro60 assay reagents, also as comparison, tested on BioFLASH instrument with QUANTA Flash Ro60 reagents
  Interventions: Device: BioCLIA Ro60
- Control Disease Samples: Samples are tested on BioCLIA Ro60 instrument with Ro60 assay reagents, also as comparison, tested on BioFLASH instrument with QUANTA Flash Ro60 reagents
  Interventions: Device: BioCLIA Ro60

INTERVENTIONS:
Device: BioCLIA Ro60 — BioCLIA Ro60 is a Chemiluminescent Immuno Assay (CLIA) as a fully automated testing process, reporting with arbitrary units, RU/mL

SUMMARY:
The study is to evaluate the clinical performance of BioCLIA Ro60 for measuring the autoantibody in autoimmune disease patients.

DETAILED DESCRIPTION:
100-200 clinically-diagnosed disease samples, as well as approximately 300 samples of various control diseases, will be used in the study. The specimen will be collected as the clinically leftover samples that have been used for routine clinical diagnosis purpose or research purpose, and with de-identification methods. Each set of samples will also be tested on a control serologic Anti-Ro60 detection kit, QUANTA Flash Ro60. Clinical sensitivity and clinical specificity will be analyzed for, also a method comparison conclusion will be drawn by comparing the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relevant diseases, including Systemic lupus erythematosus (SLE) and Sjogren's syndrome (SS)
* Or diagnosed with other control diseases, including Rheumatoid arthritis (RA), Infectious diseases and others

Exclusion Criteria:

* Treatment with medicine that submerge the autoantibody concentration to non-detectable range
* Co-diagnosed with multiple relevant diseases (e.g., SLE / SS) and/or control diseases
* Hemolyzed sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sites for clinically leftover samples accessed through Access Biologicals not confined to any demographic groups, general health status nor geographic locations
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-04-16 (Estimated); Study Completion 2020-04-16 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of BioCLIA Ro60 | 10 months
  About 500 μl or more of each de-identified sample, in the form of serum or plasma, will be tested on-board with the automated BioCLIA serologic antinuclear antibodies (ANA) assay. Result will be reported in the form or IU/ml of antibodies in the samples. Clinical sensitivity of BioCLIA Ro60 will be determined by dividing the number of Ro60 positives by the number of relevant disease samples. Clinical specificity of BioCLIA will be determined by dividing the number of Ro60 negatives by the number of control disease samples.

SECONDARY OUTCOMES:
Method comparison between BioCLIA Ro60 and BioFlash/QUANTA Flash Ro60 | 2 months
  The same samples tested in BioCLIA Ro60 will be tested on-board with the automated BioFLASH instrument with QUANTA Flash Ro60 reagents. Result will be reported in the form of CU of antibodies in the samples. Clinical sensitivity of BioFLASH/QUANTA Flash Ro60 will be determined by dividing the number of Ro60 positives by the number of relevant disease samples. Clinical specificity of BioFLASH/QUANTA Flash Ro60 will be determined by dividing the number of Ro60 negatives by the number of control disease samples. Degree of agreement between BioCLIA Ro60 and BioFLASH/QUANTA Flash Ro60 will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Chan, PhD, Principal Investigator — CRM Biotech
Locations (1):
- CRM Biotech, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No